CLINICAL TRIAL: NCT00893074
Title: The Effect of Prescription Medications in Marijuana Users
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00026278; R01DA025044 (NIH)
Record Dates: First submitted 2009-04-30; First posted 2009-05-05 (Estimated); Results first posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Marijuana Abuse
Keywords: withdrawal; acute effects; cognitive performance; Marijuana Use; Marijuana Abstinence
MeSH Terms: conditions — Marijuana Abuse; Marijuana Use | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Within-subjects cross-over evaluation of 0, 30, 60, and 120mg dronabinol per day on withdrawal, cognitive performance, and response to acute cannabis exposure
Who Masked: Participant, Outcomes Assessor
Masking Description: Dronbinol doses were double blind and placebo controlled
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0, 30, 60, and 120mg dronabinol (Other): 0, 30, 60, and 120mf dronabinol was administered in a randomized within-subjects crossover study to compare the medication dose effects of cannabis withdrawal, cognitive performance, and response to acute cannabis dosing
  Interventions: Drug: Dronabinol 30mg/day; Drug: Dronabinol 60mg/day; Drug: Dronabinol 120mg/day; Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol 30mg/day — 10mg dronabinol administered 3x/day for 5 days
  Other Names: THC; Marinol
Drug: Dronabinol 60mg/day — 20mg dronabinol administered 3x/day for 5 days
  Other Names: THC; Marinol
Drug: Dronabinol 120mg/day — 40mg dronabinol administered 3x/day for 5 days
  Other Names: THC; Marinol
Drug: Placebo — placebo dronabinol administered 3x/day for 5 days

SUMMARY:
A subset of heavy marijuana users have trouble quitting marijuana use and the number of those seeking treatment for problems related to marijuana is increasing. The purpose of this research study is to investigate whether dronabinol can reduce withdrawal effects associated with stopping marijuana use, if dronabinol can reduce the rewarding effects of smoked marijuana, and whether there are any cognitive performance deficits associated with dronabinol doses that produce such effects.

ELIGIBILITY:
Inclusion Criteria:

* current use of marijuana
* able to give informed consent

Exclusion Criteria:

* dependence on drug other than marijuana
* pregnant, breast feeding, or planning to become pregnant within the next 3 months
* currently seeking treatment for cannabis-related problems or otherwise trying to reduce use
* use of cannabis under the guidance of a physician for a medical disorder
* unstable or uncontrolled cardiovascular disease (e.g., hypertension, angina)
* allergy to study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Result] Vandrey R, Stitzer ML, Mintzer MZ, Huestis MA, Murray JA, Lee D. The dose effects of short-term dronabinol (oral THC) maintenance in daily cannabis users. Drug Alcohol Depend. 2013 Feb 1;128(1-2):64-70. doi: 10.1016/j.drugalcdep.2012.08.001. Epub 2012 Aug 22. PMID 22921474
- [Derived] Schlienz NJ, Lee DC, Stitzer ML, Vandrey R. The effect of high-dose dronabinol (oral THC) maintenance on cannabis self-administration. Drug Alcohol Depend. 2018 Jun 1;187:254-260. doi: 10.1016/j.drugalcdep.2018.02.022. Epub 2018 Apr 17. PMID 29689485
- [Derived] Lee D, Vandrey R, Mendu DR, Murray JA, Barnes AJ, Huestis MA. Oral fluid cannabinoids in chronic frequent cannabis smokers during ad libitum cannabis smoking. Drug Test Anal. 2015 Jun;7(6):494-501. doi: 10.1002/dta.1718. Epub 2014 Sep 14. PMID 25220020
- [Derived] Lee D, Vandrey R, Milman G, Bergamaschi M, Mendu DR, Murray JA, Barnes AJ, Huestis MA. Oral fluid/plasma cannabinoid ratios following controlled oral THC and smoked cannabis administration. Anal Bioanal Chem. 2013 Sep;405(23):7269-79. doi: 10.1007/s00216-013-7159-8. Epub 2013 Jul 6. PMID 23831756

RESULTS

PARTICIPANT FLOW:
Groups:
- 0, 30, 60, and 120mg Dronabinol: 0, 30, 60, and 120mg Dronabinol administered for 5 consecutive days in a double blind, placebo controlled study, with dose administered in a random order to the same study participants
Period: Overall Study
Arm/Group | 0, 30, 60, and 120mg Dronabinol
Started | 24
Completed | 13
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- Study Participant: Participants who received active drug as part of the study
Arm/Group | Study Participant
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Peak Effect of Marijuana Withdrawal
Description: Total withdrawal based on a composite score of the Marijuana Withdrawal Checklist (range 0-32; higher scores indicate greater withdrawal).
Time Frame: Day 5 of the Dronabinol abstinence period
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: 0mg daily dronabinol administered for 5 days
- 30mg Dronabinol: 30mg daily dronabinol (10mg tid) administered for 5 days
- 60mg Dronabinol: 60mg daily dronabinol (20mg tid) administered for 5 days
- 120mg Dronabinol: 120mg daily dronabinol (40mg tid) administered for 5 days
Arm/Group | Placebo | 30mg Dronabinol | 60mg Dronabinol | 120mg Dronabinol
Number analyzed (Participants) | 13 | 13 | 13 | 13
units on a scale | 4.6 (0.9) | 4.1 (0.9) | 2.9 (0.7) | 1.7 (0.4)

2. Primary Outcome: Subjective "Drug Effect" After Smoked Marijuana
Description: Subjective drug effects on a 100mm point Visual Analog Scale reported following acute cannabis dose administration during dronabinol maintenance, scale ranging 0-100, with 0 being no effect and 100 being maximum effect
Time Frame: Day 5 of the Dronabinol abstinence period
Measure: Mean (Standard Error); unit: mm of subjective drug effect
Groups:
- Placebo: Placebo dronabinol maintenance
- 30mg Dronabinol: 30mg (10mg tid) dronabinol maintenance
- 60mg Dronabinol: 60mg (20mg tid) dronabinol maintenance
- 120mg Dronabinol: 120mg (40mg tid) dronabinol maintenance
Arm/Group | Placebo | 30mg Dronabinol | 60mg Dronabinol | 120mg Dronabinol
Number analyzed (Participants) | 13 | 13 | 13 | 13
mm of subjective drug effect | 23 (3) | 28 (3) | 24 (3) | 29 (3)

3. Secondary Outcome: Heart Rate
Description: Heart rate measured after acute cannabis exposure
Time Frame: Assessed on Day 5 of dronabinol maintenance
Measure: Mean (Standard Error); unit: beats per minutes
Arm/Group | Placebo | 30mg Dronabinol | 60mg Dronabinol | 120mg Dronabinol
Number analyzed (Participants) | 13 | 13 | 13 | 13
beats per minutes | 88 (2) | 85 (2) | 80 (1) | 76 (1)

ADVERSE EVENTS:
Time Frame: 51 days
Groups:
- Placebo: Placebo maintenance
- 30mg: 30mg dronabinol maintenance
- 60mg: 60mg dronabinol maintenance
- 120mg: 120mg dronabinol maintenance
Arm/Group | Placebo | 30mg | 60mg | 120mg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 7/24 | 7/24 | 4/24 | 7/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | 30mg (N=24) | 60mg (N=24) | 120mg (N=24)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (4) | 3 (7)
Depression (Psychiatric disorders) | 5 (8) | 2 (3) | 3 (4) | 2 (4)
Dry Mouth (General disorders) | 3 (4) | 3 (5) | 3 (10) | 5 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No